CLINICAL TRIAL: NCT06267651
Title: Value Of ACE Index (Albumin, CRP And Endoscopy) In Predicting Intra Venous Steroid Response In Acute Severe Ulcerative Colitis In Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Safwat ِِِAbd elhamid eltaih, Assistant lecturer, Assiut University
Other Study IDs: Steroid in ulcerative colitis
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Early Detection of Complication of Ulcerative Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Determine if the ACE index can predict resoponse to I V steroid in Acute severe ulcerative colitis
2. identify on admission a high-risk population who may beneft from earlier second line medical treatment or surgical intervention. ( steroid non responder groups )

DETAILED DESCRIPTION:
UlCerative colitis is characterized by mucosal inflammation initiating in the rectum and extending proximally in the colon in a continuous fashion. In patients with acute severe colitis, prompt hospital admission is required, A multidisciplinary approach is fundamental, and contacting a colorectal surgeon at the moment of admission is recommended. Sometimes, emergency surgery might be required early on in case of toxic megacolon, perforation or massive bleeding.

Although treatment initiation should not be postponed in severe cases, excluding differential diagnoses, including C. difficile infection, is crucial. A limited flexible sigmoidoscopy without bowel preparation should be performed to assess disease severity .(1) aggressive medical therapy, starting with intravenous corticosteroids. Intravenous [IV] steroids remain the frst-line medical therapy for patients admitted with acute severe UC [ASUC], as defned by Truelove and Witts criteria,)(2) Almost one-third of patients, however, may not respond to IV steroids and go on to require second-line medical therapies [primarily inﬂiximab or ciclosporin] or a colectomy .

A signifcant body of research in recent years has focused on predicting outcome in patients with ASUC treated with IV steroids; ,(3) In 2022 the novel ACE was reported [Albumin, CRP, and Endoscopy] Index in acute colitis, which used biochemical and endoscopic parameters to predict steroid non-response on admission (albumin ≤ 30g/L [0 or 1] + C-reactive protein [CRP] ≥ 50 mg/L [0 or 1] + endoscopically severe according to physician's global assessment component of the Mayo score [0 or 1]), We can identify a high-risk subset of patients for targeted counselling and early administration of second-line therapy; this is particularly crucial as treatment delays are associated with increased mortality.

ELIGIBILITY:
Inclusion Criteria:

- Adult Patients (≥18 years) known ulcerative colitis presented with activity .

2- newly diagnosed ulcerative colitis

Exclusion Criteria:

* 1) patient presented with CMV colitis 2) Clostridium difficile infection 3) Elective admission

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Pt above 18 years old presented with Acute severe ulcerative colitis treated by Iv steroid
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Early prevention of complication of ulcerative colitis | 2 years
  Histopathology of colon biopsy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santos AL, Lopes S, Peixoto A, Garrido I, Medas R, Andrade P, Macedo G. The ACE (Albumin, CRP, and Endoscopy) Index in Acute Colitis: Simplify to a Better Prognostic Prediction. Inflamm Bowel Dis. 2021 Oct 20;27(11):e140. doi: 10.1093/ibd/izab189. No abstract available. PMID 34331454